CLINICAL TRIAL: NCT05968846
Title: Repeat PET/CT Imaging of Patients With Systemic Amyloidosis Using Amyloid Reactive Peptide 124I-AT-01 (124I-p5+14, Iodine-124I-evuzamitide) to Measure Changes in Organ-specific Amyloid Load
Brief Title: Repeat PET/CT Imaging of Patients With Amyloid 124I-AT-01 to Measure Changes in Organ-specific Amyloid Load
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UTMC-AT01-163117
Record Dates: First submitted 2023-06-30; First posted 2023-08-01 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Systemic Amyloidosis
Keywords: systemic amyoidosis; p5+14; AT-01; PET/CT; evuzamitide
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Iodine-124

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients will receive a single IV injection of 124I-AT-01 radiotracer and PET/CT imaging (Experimental): 124I-AT-01 (124I-p5+14, iodine-124I evuzamitide) is an iodine-124 (124I) labeled 45 L-amino acid peptide suitable for PET/CT imaging. The peptide binds many forms of amyloid through multivalent electrostatic interactions with the amyloid fibril and ubiquitous heparan sulfate proteoglycans.
  124I-AT-01 has been evaluated previously in an open-label Phase 1/2 clinical trial, AMY1001, performed at the University of Tennessee Medical Center (IND# 132282; NCT T03678259).
  In this repeat imaging study, patients previously enrolled in the AMY1001 study, in whom positive PET/CT imaging findings were observed will undergo repeat imaging to assess changes in radiotracer uptake in the liver, spleen, heart and kidneys.
  Interventions: Drug: Injection of peptide p5+14 radiolabeled with iodine-124 (124I-AT-01)

INTERVENTIONS:
Drug: Injection of peptide p5+14 radiolabeled with iodine-124 (124I-AT-01) — 124I-AT-01 (124I-p5+14, iodine-124I evuzamitide) is a a novel iodine-124 (124I) labeled 45 L-amino acid peptide suitable for PET/CT imaging that has been shown to bind systemic amyloid deposits of diverse types in all organs, including the heart. The peptide binds amyloid through multivalent electrostatic interactions with the amyloid fibril and ubiquitous heparan sulfate proteoglycans.
  Other Names: 124I-p5+14; iodine-124-evuzamitide

SUMMARY:
The goal of this research study is to determine whether changes in organ-specific uptake of 124I- AT-01 can be measured by PET/CT imaging and further, whether these values correlate with changes in a subject's disease status and thereby enable monitoring of disease response over time in terms of organ-specific amyloid load.

DETAILED DESCRIPTION:
This is a single center, open label, prospective study using 124I-AT-01 PET/CT imaging to evaluate changes in amyloid load in patients with systemic amyloidosis who had undergone 124I-AT-01 imaging.

Consented eligible patients will provide 3 tablespoons of blood for the following laboratory tests: CMP, CBC, CRP, Troponin, NT-proBNP, LDH, FLC and anti-drug antibody (ADA) analyses. A urine sample will also be collected to assess renal function. If required, a pregnancy test will be administered.

Patients will then undergo a transthoracic echocardiographic examination and vital sign assessment before receiving an intravenous injection of no more than 2 mCi 124I-AT-01 followed, 5 h thereafter, by repeat vital sign measurements and PET/CT imaging from crown to thighs with a dynamic PET acquisition over the heart. Previously acquired 124I- AT-01 PET/CT images will be used as baseline values to determine quantitative changes in uptake of the radiotracer in the heart, liver, spleen, and kidney (and other organs deemed positive following visual inspection of the baseline and repeat imaging) as a measure of changes in amyloid load. Optionally, if the patients can return to the study site within ~30 days post injection of 124I-AT-01, a second (post-injection) blood draw and ADA evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements.
* Must have a diagnosis of systemic amyloidosis based on the patient's medical record.
* Must have undergone PET/CT imaging with 124I-AT-01 as part of the AMY1001 study (IND #132282) with visually positive uptake of radiotracer in at least one abdominothoracic organ.
* Must have been imaged with 124I-AT-01 as part of the AMY1001 study (IND #132282) more than 12 months prior to repeat imaging.
* Females: must be non-pregnant and non-lactating and either: surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy); post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the laboratory involved).

Exclusion Criteria:

* Disabling dementia or other mental or behavioral disease.
* Patients on dialysis.
* Inability or unwillingness to comply with the study requirements.
* Patients taking heparin, or heparin derivatives (e.g. low molecular weight heparins) for anticoagulation.
* Other reason that would make the subject inappropriate for entry into this study.
* Inability to lie still for 60 minutes on the PET/CT scanner.
* History of iodine (potassium iodide) allergy.
* Positive ADA finding defined as significantly higher than normal human serum mean values AND with a mean value at least five times greater than the mean value of the normal human serum control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
To measure visual and quantitative changes in organ-specific uptake of 124I-AT-01 | From enrollment to the end of the study is 8 days
  The goal of this research study is to determine whether changes in organ-specific uptake of 124I- AT-01 can be measured by PET/CT imaging and further, whether these values correlate with changes in a subject's disease status and thereby enable monitoring of disease response over time in terms of organ-specific amyloid load. The specific aim of this study is to measure visual and quantitative changes in organ-specific uptake of 124I-AT-01 from baseline, in patients with systemic amyloidosis, using PET/CT imaging.

OTHER OUTCOMES:
Measures of Interest | From enrollment to the end of the study is 8 days
  For AL, ATTR and all patients, we will correlate visual and quantitative changes in 124I- AT-01 uptake, from baseline, in the heart, liver and kidney with echocardiographic parameters (including left ventricular wall thickness (cm), intraventricular wall thickness (cm), and global logitudinal strain (%)) and serum biomarker levels (including NTproBNP, eGFR, creatinine, AST and ALT) assessed prior to imaging and from data recorded in the patients' medical record.
Measure of Interest | From enrollment to the end of the study is 8 days
  For AL, ATTR and all patients, we will correlate visual and quantitative changes in organ-specific 124I-AT-01 uptake (percent change in radiotracer uptake from baseline) with change in disease status (progression, response, or stable state) when this can be established from data (serum biomarkers and cardiac imaging parameters) in the patients' medical record or collected during the AMY1001 trial.
Measure of Interest | From enrollment to the end of the study is 8 days
  For all patients, correlate organ-specific percent change in radiotracer uptake with type of therapeutic intervention and assess qualitatively whether the patient feels that their disease is improving or worsening.
Measure of interest | From enrollment to the end of is the study is 8 days
  For AL patients, correlate visual and quantitative changes in organ-specific 124I-AT-01 uptake (percent change in radiotracer uptake from baseline) with change in serum free light chains over the period between imaging studies, when available in the medical record.
Measure of Interest | From enrollment to the end of the study is 8 days
  Compare changes, when possible, in radiotracer distribution from baseline based on analysis dynamic PET data.
Measure of Interest | From enrollment to the end of the study is 8 days
  Compare changes, when possible, in ejection fraction from baseline based on analysis dynamic PET data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Graduate School of Medicine, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No